CLINICAL TRIAL: NCT03607669
Title: Manganese-Enhanced Magnetic Resonance Imaging: Applications in Cardiomyopathy
Brief Title: Manganese-Enhanced Magnetic Resonance Imaging of the Myocardium
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC16109
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Cardiomyopathy; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Controls: Healthy volunteers of similar age and gender
  Interventions: Other: Mangafodipir trisodium
- Ischaemic Cardiomyopathy: Patients with ischaemic cardiomyopathy and NYHA II-III heart failure
  Interventions: Other: Mangafodipir trisodium
- Hypertrophic Cardiomyopathy: Patients with hypertrophic cardiomyopathy and NYHA II-III heart failure
  Interventions: Other: Mangafodipir trisodium
- Dilated Cardiomyopathy: Patients with dilated cardiomyopathy and NYHA II-III heart failure
  Interventions: Other: Mangafodipir trisodium

INTERVENTIONS:
Other: Mangafodipir trisodium — Manganese-based MRI contrast agent

SUMMARY:
Scanning the heart using magnetic resonance imaging (MRI) enables detailed assessment of its structure and function. MRI can give more detailed information about the heart by using a contrast 'dye' that is injected into a vein during the scan. This can highlight abnormal areas within the heart. Current contrast dyes help identify scarring within the heart, which is useful in people who have had heart attacks. The investigators plan to test new contrast dye containing manganese, which works differently to current agents. They believe it will provide unique insight into how the heart works.

There are many different causes of heart problems and the investigators plan to use this new contrast agent to scan three patient groups; (i) heart disease caused by heart attacks, (ii) heart disease with abnormal thickening of the heart muscle, and (iii) heart disease where the heart becomes stretched and enlarged. Healthy volunteers will be scanned for comparison.

The study will be carried out at the Royal Infirmary of Edinburgh. Adults between 18 and 65 with stable heart failure can be considered. Women who may be pregnant are unable to participate, as is anyone who has some types of metal in their body, as these people can't have an MRI scan safely. All participants will have 2 MRI scans lasting about an hour each, at least 2 days apart. Some participants will be have 4 MRI scans, over a longer time period. The investigators will also take some blood samples and record a tracing of the heart rhythm and will ensure there are no abnormal side-effects by telephone follow up.

The investigators believe this new agent has potential to better measure disease in the heart, improve the ability to establish the cause of heart disease and help monitor the disease over time as well as guide future treatment for individual patients.

ELIGIBILITY:
Inclusion Criteria:

All subjects to be entered must:

* ≥ 18 years of age
* if female, be non-pregnant as evidenced by a urine pregnancy test or post-menopausal or surgically sterile
* provide written informed consent after having received oral and written information about the study

Additionally, cohort-specific inclusion criteria as follows:

Healthy Volunteers

• Healthy adult with no known pre-existing medical conditions

Ischaemic Cardiomyopathy

* Ischaemic cardiomyopathy as diagnosed by reduced LV ejection fraction (≤40%) secondary to one or more ischaemic events
* Angiographically demonstrated LMS, LAD disease, or ≥2 vessel disease
* NHYA class I-III heart failure, with stable symptoms not requiring change to diuretic therapy in the preceding month

Dilated Cardiomyopathy

* Dilated cardiomyopathy characterised with echocardiography by reduced left ventricular systolic function with impaired systolic function (ejection fraction <40%).
* NHYA class I-III heart failure, with stable symptoms not requiring change to diuretic therapy in the preceding month

Hypertrophic Cardiomyopathy

* Established diagnosis of hypertrophic cardiomyopathy
* Left ventricular wall thickness ≥15mm in any segment
* Repolarisation abnormalities on 12-lead electrocardiogram NHYA class I-III heart failure, with stable symptoms not requiring change to diuretic therapy in the preceding month

Exclusion Criteria:

* have a positive pregnancy test
* women who are breast feeding
* received an investigational drug or device within 30 days prior to administration of Mangafodipir
* have known hypersensitivity to ondansetron or other selective serotonin 5-HT3 receptor blockers
* have a history of ongoing drug abuse or alcoholism
* have a history of torsades or prolonged QT/QTc interval
* atrioventricular block (1st, 2nd or 3rd degree)
* atrial fibrillation or flutter
* have NYHA Grade IV heart failure
* have abnormal liver function tests or a history of liver disease
* have a baseline eGFR (estimated glomerular filtration rate) of <30 mL/min)
* have uncontrolled hypertension
* have any contraindications to MRI, including implanted devices/pacemakers
* be maintained on either a calcium channel blocker or digoxin
* known diagnosis of phaeochromocytoma

Additionally, cohort-specific exclusion criteria as follows:

Hypertrophic Cardiomyopathy

* Coronary artery stenosis >50% any vessel
* Previous myocardial infarction
* Previous alcohol septal ablation
* Moderate or severe aortic stenosis (mean gradient >25 mmHg, mean AVA ≤1.5 cm2 or peak velocity ≥3 m/sec),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Edinburgh Heart Centre will be invited to participate. Inpatients and outpatients are eligible. Healthy volunteers will be invited to participate by local recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Myocardial calcium-handling | 1 year
  Quantification of myocardial calcium handling by T1 mapping, in healthy controls, and patient groups.

SECONDARY OUTCOMES:
Myocardial infarction quantification | 1 year
  Quantification of infarct size using manganese, and comparison with Gadolinium enhanced MRI.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD PhD, Study Director — University of Edinburgh
Locations (1):
- Queen's Medical Research Institute, University of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spath NB, Singh T, Papanastasiou G, Baker A, Janiczek RJ, McCann GP, Dweck MR, Kershaw L, Newby DE, Semple S. Assessment of stunned and viable myocardium using manganese-enhanced MRI. Open Heart. 2021 Jun;8(1):e001646. doi: 10.1136/openhrt-2021-001646. PMID 34099530